CLINICAL TRIAL: NCT01804933
Title: Influence of Profound Muscle Relaxation on Muscle Trauma and Postoperative Pulmonary Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ying Xiao (Other)
Responsible Party: Sponsor-Investigator, Ying Xiao, Associate Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 伦审[2012]326号
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Profound Muscle Relaxation; Muscle Trauma; Postoperative Analgesic Demand; Postoperative Pulmonary Function
Keywords: profound muscle relaxation; muscle trauma; postoperative analgesic demand; postoperative pulmonary function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- conventional neuromuscular blockade (No Intervention): No rocuronium will be administered intraoperatively unless there is surgeons' complain or patients movement
- optimal neuromuscular blockade (Active Comparator): Rocuronium dose will be infused to maintain depth of NMB at TOF count 1 intraoperatively
  Interventions: Drug: profound neuromuscular blockade
- profound neuromuscular blockade (Experimental): Rocuronium dose will be infused to maintain a depth of NMB to PTC 1~2 intraoperatively
  Interventions: Drug: profound neuromuscular blockade

INTERVENTIONS:
Drug: profound neuromuscular blockade — Rocuronium dose will be infused to maintain a depth of NMB to PTC 1~2 intraoperatively
  Arms: optimal neuromuscular blockade; profound neuromuscular blockade

SUMMARY:
Although deep anesthesia can produce skeleton muscle relaxation,unnecessary deep anesthesia often had adverse cardiac effects and was related to 2-year mortality in cancer patients.The use of muscle relaxants allowed the depth of anesthesia to be optimized.However, for many anesthesiologists,in fear of residual postoperative neuromuscular blockade,intraoprative administration of muscle relaxants had to be minimized in spite of poor surgical conditions.

This study, however, is designed to test the hypothesis that profound neuromusclular blockade reduces muscle trauma caused by self-retaining retractor and thus cut down postoperative analgesic requirement.On the other hand,profound muscle relaxation can decrease postoperative diaphragmatic dysfunction and abdominal muscle trauma, which can improve postoperative pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1~2,scheduled to undergo upper abdominal surgery by midline incision

Exclusion Criteria:

* neuromuscular disorder
* history of malignant hyperthemia
* allergy to medications used during general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
degree of muscle trauma | 72h postoperatively
  serum CK

SECONDARY OUTCOMES:
postoperative analgesic requirement | 7days postoperatively
  consumption of morphine

OTHER OUTCOMES:
postoperaive pulmonary function | 3days postoperatively
  FEV1 FVC PEF

CONTACTS AND LOCATIONS:
Overall Officials: Ying Xiao, MD, PhD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China